CLINICAL TRIAL: NCT01005823
Title: A Safety, Tolerability and Pharmacokinetic Study of LEO 29102 in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 29102-C03; EudraCT No. 2009-014303-30
Record Dates: First submitted 2009-10-23; First posted 2009-11-02 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2010-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LEO 29102 cream 0.3 mg/g (Active Comparator)
  Interventions: Drug: LEO 29102 cream
- LEO 29102 cream 1.0 mg/g (Active Comparator)
  Interventions: Drug: LEO 29102 cream
- LEO 29102 cream 2.5 mg/g (Active Comparator)
  Interventions: Drug: LEO 29102 cream
- LEO 29102 placebo cream (Placebo Comparator)
  Interventions: Drug: LEO 29102 placebo cream

INTERVENTIONS:
Drug: LEO 29102 cream — Twice daily application for 7 days
  Arms: LEO 29102 cream 0.3 mg/g; LEO 29102 cream 1.0 mg/g; LEO 29102 cream 2.5 mg/g
Drug: LEO 29102 placebo cream — LEO 29102 placebo cream
  Arms: LEO 29102 placebo cream

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of 7 days treatment with LEO 29102 in adult patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55 years
* Atopic dermatitis of 850-1700cm2
* In good health

Criteria for exclusion:

* Co-morbid conditions
* Hepatic dysfunction
* Clinical infection
* Immunocompromised status
* Clinically significant illness
* Use of immunomodulating treatment
* Medications related to respiratory system or to heart rhythm

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory testing, ECG, vital signs | Day 9

SECONDARY OUTCOMES:
To assess the efficacy of LEO 29102 cream in the treatment of AD | Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Kahlid Aboufarha, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA International, University Medical Centre, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No